CLINICAL TRIAL: NCT00882674
Title: An Exploratory Study to Evaluate the Biological Activity of R1507, a Human Monoclonal Antibody Antagonist of the Insulin-like Growth Factor Receptor (IGF-1R) in Women With Operable Breast Cancer
Brief Title: A Study to Evaluate the Biological Activity of R1507 in Women With Operable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NP22002; 2008-004128-22
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — RG-1507 monoclonal antibody

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG1507

INTERVENTIONS:
Drug: RG1507 — 16mg/kg, 9mg/kg, 3mg/kg or 1mg/kg iv on Day 1 in one of 4 cohorts of patients

SUMMARY:
This 2 part study will explore the pharmacodynamic effects of R1507 in breast cancer tumor cells in female patients with operable breast cancer. In the first part of the study, patients will receive a single dose of R1507, 16mg/kg iv, on day 1; pre-and post-treatment (at breast surgery on day 8) breast tissue samples will be obtained for measurement of IGF-1R expression. If sufficient biological activity is demonstrated, 3 additional cohorts of patients will be entered into Part 2 of the study, to receive a single dose of 9mg, 3mg/kg or 1mg/kg iv R1507, respectively. The anticipated time on study treatment is < 3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* invasive, and operable, breast cancer;
* ECOG Performance Status of 0 or 1.

Exclusion Criteria:

* evidence of metastatic disease;
* inflammatory breast cancer;
* prior hormonal or systemic therapy for breast cancer;
* prior treatment with an agent targetting the IGF-1R pathway;
* patients receiving concurrent radiotherapy, or who have received radiotherapy within 28 days prior to receipt of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in IGF-1R expression | From initial diagnosis to tumor excision

SECONDARY OUTCOMES:
Correlation of R1507 pharmacokinetic parameters with biological changes in tumor tissue | Days 1, 8 and 31
Adverse events, laboratory parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Edinburgh, United Kingdom